CLINICAL TRIAL: NCT00320996
Title: SGO Society of Gynecologic Oncologists Data Outcomes Project
Status: Terminated | Type: Observational
Why Stopped: This is not a clinical trial and was entered in the system in error.
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Other Study IDs: 3002C
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Pelvic Tumor
Keywords: Pelvic mass
MeSH Terms: conditions — Pelvic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
SGO Society of Gynecologic Oncologists Data Outcomes Project.

DETAILED DESCRIPTION:
Examines data over period of time

ELIGIBILITY:
Inclusion Criteria:

1. Must have a pelvic mass with surgery taking place.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Females with a pelvic mass who will have surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2002-03 (Actual); Primary Completion 2004-07 (Actual); Study Completion 2005-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harriet Smith, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States